CLINICAL TRIAL: NCT00747513
Title: A Multi-component Program to Improve Lifestyle Habits and Reduce Obesity in Children
Brief Title: A Multi-component Program to Reduce Obesity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Rashi Foundation (Other); D-Cure, Israel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA- 08-5401-LL-CTIL
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Obesity
Keywords: school; prevention; overweight; children; diet; physical activity; fitness
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): intervention group
  Interventions: Behavioral: lifestyle program

INTERVENTIONS:
Behavioral: lifestyle program — a comprehensive program designed to encourage healthier food choices and eating habits and increased physical activity among children, by use of school, family and community measures.

SUMMARY:
In an attempt to challenge the increasing prevalence of childhood obesity, many programs have been executed in order to improve childrens' lifestyle. Programs involved either school, family or environmental measures. In most, success was only limited.

The purpose of this trial is to examine the ability of a low-cost multi-component program to improve behavioral, diet and activity habits in both school, family and afternoon settings. Ths ultimate goal is to construct and assess a lifestyle modification program that can be implemented in schools and kindergartens on a national level.

Participants will be ~2,500 children aged 5-12 from 22 kindergartens and elementary schools, divided into control and intervention centers.

Teachers and students will be provided with materials in order to perform activities on healthy food and drink choices and habits during the school day. Schools will offer increased physical activity opportunities to children, as will afternoon community centers. Children will be given personal exercise items. Parents will be offered lectures on topics of diet and activity. Diet and activity habits will be assessed by a questionnaire, and height, weight and body fat percentage will be measured before and after the program.

ELIGIBILITY:
Inclusion Criteria:

* schools with lunch served
* school principal agreement
* school has 2 weekly PE classes
* parent and children consent given

Exclusion Criteria:

* consent not given

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3600 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
screen time | 12 months
physical activity | 12 months
breakfast consumption | 12 months
eating family meals | 12 months
number of fruits and vegetables eaten per day | 12 months
drinking water | 12 months
body mass index | 12 months

SECONDARY OUTCOMES:
body fat percentage | 12 months
daily dairy product intake | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Liat Lerner-geva, MD PhD, Principal Investigator — Women and Children's Health Research Unit, Gertner Institute, Tel Hashomer, Israel
Locations (22):
- Israel (22):
  - El Biader, Hura
  - El Magad, Hura
  - Harel Elementary School, Lod
  - Mabuim School, Merhavim
  - Merhavim School, Merhavim
  - Rothchild School, Or Akiva
  - Amirim School, Qiryat Yam
  - Miflasim School, Qiryat Yam
  - El Gazali, Rahat
  - Omar El Hatab, Rahat
  - Achva School, Ramla
  - Sharet Elementary School, Ramla
  - Fikus Preschool, Rosh HaAyin
  - Ilanot Preschol, Rosh HaAyin
  - Kinor Preschool, Rosh HaAyin
  - Meitar Preschool, Rosh HaAyin
  - Nevel Preschool, Rosh HaAyin
  - Teena Preschool, Rosh HaAyin
  - Maimon School, Shlomi
  - Hassan Arafe School, Tel Aviv
  - Lev Yafo School, Tel Aviv
  - Noam School, Tiberias